CLINICAL TRIAL: NCT04436198
Title: The Investigation of Capsular Tension Rings in Intraocular Lens Rotation
Brief Title: Capsular Tension Rings in Intraocular Lens Rotation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no longer feasible
Sponsor: Rachel Lieberman (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Rachel Lieberman, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20200112H
Record Dates: First submitted 2020-05-19; First posted 2020-06-17 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Cataract; Ophthalmoplegia; Ophthalmologic Complication
Keywords: ophthalmology; capsular tension ring; rotation
MeSH Terms: conditions — Cataract; Ophthalmoplegia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment group: toric IOL plus capsular tension ring (Experimental)
  Interventions: Device: MORCHER® EYEJET® CTR Types 14, 14A, and 14C
- Control group: toric IOL only (Active Comparator)
  Interventions: Device: Toric IOL Only

INTERVENTIONS:
Device: MORCHER® EYEJET® CTR Types 14, 14A, and 14C — Intervention. Toric IOL + CTR. Whether the subject receives 14, 14A, or 14C is an either or scenario depending on the eye's axial length and is a single intervention:
  Axial length > 28.0 mm: CTR model 14A Axial length 24.0-28.0 mm: CTR model 14C Axial length < 24.0 mm: CTR model 14
  Lens Selection: The patients will undergo standard of care preoperative measurements and planning. The surgeon will evaluate preoperative measurements and use lens calculations, as well as a discussion with the patient, to identify whether a toric lens will be used and to determine the IOL power, cylinder, and target axis (standard of care). Preoperative measurements will be taken using IOL-Master 700, with the addition of the Pentacam and automatic keratometry as needed (standard of care). The toric lens used will be the TECNIS IOL. It will be used on label (standard of care).
  Arms: Treatment group: toric IOL plus capsular tension ring
Device: Toric IOL Only — Control. Toric IOL only. Standard of care cataract surgery without placement of a capsular tension ring.
  Lens Selection: The patients will undergo standard of care preoperative measurements and planning. The surgeon will evaluate preoperative measurements and use lens calculations, as well as a discussion with the patient, to identify whether a toric lens will be used and to determine the IOL power, cylinder, and target axis (standard of care). Preoperative measurements will be taken using IOL-Master 700, with the addition of the Pentacam and automatic keratometry as needed (standard of care). The toric lens used will be the TECNIS IOL. It will be used on label (standard of care).
  Arms: Control group: toric IOL only

SUMMARY:
To investigate whether implantation of a capsular tension ring device will affect the degree of rotation of an implanted toric intraocular lens following cataract surgery.

DETAILED DESCRIPTION:
The study is a prospective, subject-blinded investigation of whether implanting capsular tension rings with intraocular lenses affects rotational stability of the lens.

Lens Selection: The patients will undergo standard of care preoperative measurements and planning. The surgeon will evaluate preoperative measurements and use lens calculations, as well as a discussion with the patient, to identify whether a toric lens will be used and to determine the IOL power, cylinder, and target axis (standard of care). Preoperative measurements will be taken using IOL-Master 700, with the addition of the Pentacam and automatic keratometry as needed (standard of care). The toric lens used will be the TECNIS IOL. It will be used on label (standard of care).

Randomization: Each eye undergoing cataract surgery will be randomized into a control or treatment group. If both eyes meet enrollment criteria, then each eye will be randomized independently.

* Control group: toric IOL only
* Treatment group: toric IOL plus capsular tension ring

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active duty and DoD beneficiaries aged 30 years or older undergoing cataract surgery
* Corneal astigmatism ≥ 1.0 D and a surgical plan that includes a toric intraocular lens for astigmatism correction. (The lens used will be the TECNIS IOL. It will be used on label)
* No observed zonular or capsular problems prior to, or at the time of, capsular tension ring insertion

Exclusion Criteria:

* Patients undergoing cataract surgery who do not have corneal astigmatism ≥1.0 D.
* Any observed zonular or capsular problems prior to, or at the time of, capsular tension ring insertion.
* Pre-existing ocular conditions, including:Pre-existing ocular conditions, including:

  * Pseudoexfoliation syndrome in one or both eyes
  * Prior incisional ocular surgery
  * Lens subluxation
  * Poor dilation or inability to position at the slit lamp (making postoperative outcome measurements difficult or impossible)
  * Plans for extensive travel or to move away during the postoperative evaluation period
  * Other conditions that would influence the capsule or lens positioning
* Surgical plan to include other procedures at the time of initial cataract surgery, such as Limbal Relaxing Incisions (LRIs), Micro-Incisional Glaucoma Surgery (MIGS), etc.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Lieberman, MD, Principal Investigator — United States Air Force
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] Novis C. Astigmatism and toric intraocular lenses. Curr Opin Ophthalmol. 2000 Feb;11(1):47-50. doi: 10.1097/00055735-200002000-00007. PMID 10724827
- [Background] Shimizu K, Misawa A, Suzuki Y. Toric intraocular lenses: correcting astigmatism while controlling axis shift. J Cataract Refract Surg. 1994 Sep;20(5):523-6. doi: 10.1016/s0886-3350(13)80232-5. PMID 7996408
- [Background] Holland E, Lane S, Horn JD, Ernest P, Arleo R, Miller KM. The AcrySof Toric intraocular lens in subjects with cataracts and corneal astigmatism: a randomized, subject-masked, parallel-group, 1-year study. Ophthalmology. 2010 Nov;117(11):2104-11. doi: 10.1016/j.ophtha.2010.07.033. Epub 2010 Sep 16. PMID 20846724
- [Background] Felipe A, Artigas JM, Diez-Ajenjo A, Garcia-Domene C, Alcocer P. Residual astigmatism produced by toric intraocular lens rotation. J Cataract Refract Surg. 2011 Oct;37(10):1895-901. doi: 10.1016/j.jcrs.2011.04.036. Epub 2011 Aug 23. PMID 21865007
- [Background] Rastogi A, Khanam S, Goel Y; Kamlesh; Thacker P, Kumar P. Comparative evaluation of rotational stability and visual outcome of toric intraocular lenses with and without a capsular tension ring. Indian J Ophthalmol. 2018 Mar;66(3):411-415. doi: 10.4103/ijo.IJO_875_17. PMID 29480253
- [Background] Shah GD, Praveen MR, Vasavada AR, Vasavada VA, Rampal G, Shastry LR. Rotational stability of a toric intraocular lens: influence of axial length and alignment in the capsular bag. J Cataract Refract Surg. 2012 Jan;38(1):54-9. doi: 10.1016/j.jcrs.2011.08.028. Epub 2011 Nov 4. PMID 22055077
- [Background] Zhao Y, Li J, Yang K, Li X, Zhu S. Combined Special Capsular Tension Ring and Toric IOL Implantation for Management of Astigmatism and High Axial Myopia with Cataracts. Semin Ophthalmol. 2018;33(3):389-394. doi: 10.1080/08820538.2016.1247181. Epub 2016 Dec 22. PMID 28005433
- [Background] Safran SG. Use of Capsular Tension Ring to Prevent Early Post-operative Rotation of a Toric Intraocular Lens in High Axial Myopia. JCRS Online Case reports. 2015.
- [Background] Sagiv O, Sachs D. Rotation stability of a toric intraocular lens with a second capsular tension ring. J Cataract Refract Surg. 2015 May;41(5):1098-9. doi: 10.1016/j.jcrs.2015.04.004. Epub 2015 Apr 28. PMID 25937341
- [Background] Jung NY, Lim DH, Hwang SS, Hyun J, Chung TY. Comparison of clinical outcomes of toric intraocular lens, Precizon vs Tecnis: a single center randomized controlled trial. BMC Ophthalmol. 2018 Nov 9;18(1):292. doi: 10.1186/s12886-018-0955-3. PMID 30413154

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Treatment Group: Toric IOL Plus Capsular Tension Ring | Control Group: Toric IOL Only
Started (A single participant contributed 1 eye to treatment group and 1 eye to control group and is therefore double counted. There were actually 12 participants, not 13.) | 7; 7 eyes | 6; 6 eyes
Completed | 5; 5 eyes | 3; 3 eyes
Not Completed | 2; 2 eyes | 3; 3 eyes

BASELINE CHARACTERISTICS:
Population: There were 12 participants, with one single participant contributing 1 eye to control and 1 eye to treatment. The participant is therefore double counted as they have an eye in control and an eye in treatment. Total has been adjusted to reflect that there were 12 participants total even though 13 were calculated due to the calculator calculating eyes as units, not participants as units.
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group: Toric IOL Plus Capsular Tension Ring | Control Group: Toric IOL Only | Total
Number analyzed (Participants) | 7 | 6 | 12
Number analyzed (eyes) | 7 | 6 | 13
Age, Categorical [Count of Units; unit: eyes] — Population: As this study measured eyes not subjects, one subject had an eye in control and the other eye in treatment. As such, row population is larger than overall population as one subject is reported in both rows.
  eyes
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 1 | 1
    >=65 years | 7 | 5 | 12
Sex: Female, Male [Count of Units; unit: eyes] — Population: As this study measured eyes not subjects, one subject had an eye in control and the other eye in treatment. As such, row population is larger than overall population as one subject is reported in both rows.
  eyes
    Female | 5 | 3 | 8
    Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Units; unit: eyes] — Population: As this study measured eyes not subjects, one subject had an eye in control and the other eye in treatment. As such, row population is larger than overall population as one subject is reported in both rows.
  eyes
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 1 | 0 | 1
    White | 4 | 3 | 7
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: eyes] — Population: As this study measured eyes not subjects, one subject had an eye in control and the other eye in treatment. As such, row population is larger than overall population as one subject is reported in both rows.
  eyes
    United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Degree of Toric Rotation Away From Target Axis in Enrolled Eye/s
Description: The eye(s) enrolled in the study will be dilated and slit lamp photography taken using retroillumination.
  The capsular tension ring will not be visible in the slit lamp photos or during the eye exams. The patient will be blinded as to which eye is in the treatment or control group. The slit lamp photos will be de-identified and used to determine the axis of the toric IOL by evaluators blinded to the patient identity and control/treatment group. The toric axis will be identified using either ImageJ (NIH) or Adobe Illustrator by measuring the angle between a straight line drawn across the toric axis markers and a straight line at the horizontal axis (0 degrees).
Time Frame: 6 months
Measure: Mean (Full Range); unit: degree of rotation
Units Other Than Participants: eyes
Arm/Group | Treatment Group: Toric IOL Plus Capsular Tension Ring | Control Group: Toric IOL Only
Number analyzed (Participants) | 5 | 3
Number analyzed (eyes) | 5 | 3
degree of rotation
  average difference between intended toric axis (degrees) | 5.739 [.506 to 11.383] | 3 [2.82 to 15.5173]
  average difference between intended axis (degrees) | 5 [1 to 13] | 10 [7 to 13]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment Group: Toric IOL Plus Capsular Tension Ring | Control Group: Toric IOL Only
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT04436198/Prot_SAP_000.pdf